CLINICAL TRIAL: NCT01984554
Title: Observational Study on the Use of IV (Intravenous) Iron Therapy Among Subjects With Iron Deficiency Anemia
Status: Completed | Type: Observational
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1VIT13033
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Iron Deficiency Anemia (IDA)
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Ferric Carboxymaltose (FCM): Dosing levels, treatment choice, number and scheduling of infusions are all at the discretion of the subject and the subject's prescribing physician.
- Iron Sucrose: Dosing levels, treatment choice, number and scheduling of infusions are all at the discretion of the subject and the subject's prescribing physician
- Iron Dextran: Dosing levels, treatment choice, number and scheduling of infusions are all at the discretion of the subject and the subject's prescribing physician
- Ferumoxytol: Dosing levels, treatment choice, number and scheduling of infusions are all at the discretion of the subject and the subject's prescribing physician

SUMMARY:
The primary objective of this study is to compare the total costs to sites and payers of administering IV iron over the 30-day observation period for subjects with IDA who receive Ferric Carboxymaltose (FCM) relative to those who receive iron sucrose, iron dextran, and ferumoxytol.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the total costs to sites and payers of administering IV iron over the 30-day observation period for subjects with IDA who receive Ferric Carboxymaltose (FCM) relative to those who receive iron sucrose, iron dextran, and ferumoxytol.

ELIGIBILITY:
Inclusion Criteria:

* Must present for the first dose of a current cycle of IV treatment for IDA
* Must be over 18 years of age
* Must be willing and able to provide informed consent, including permission to obtain information from their medical records.
* Must be able to read and understand English.

Exclusion Criteria:

* Subjects not diagnosed with IDA.
* Subjects requiring more than one treatment cycle within 30 days.
* Subjects receiving maintenance IV iron therapy.
* Subjects treated with IV iron within the 30-day period prior to study enrollment.
* Subjects who received investigational medication in the six months prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting for IDA treatment
Sampling Method: Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Site costs of administering IV iron to subjects to be assessed by applying unit costs to information collected directly on the eCRF (electronic Case Report Form). | 30 day observation period

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States